CLINICAL TRIAL: NCT05304273
Title: COMPARATIVE STUDY OF EFFECTS BETWEEN LETROZOLE PLUS MISOPROSTOL AND MIFEPRISTONE PLUS MISOPROSTOL IN TERMINATING NON-VIABLE FIRST TRIMESTER PREGNANCIES
Brief Title: Comparison Between Letrozole and Mifepristone in Medical Termination of First Trimester Miscarriages
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Calcutta National Medical College and Hospital (Other Government)
Responsible Party: Principal Investigator, Dr.Jhuma Biswas, Associate Professor, Dept. of Obstetrics and Gynecology, Calcutta National Medical College and Hospital, Calcutta National Medical College and Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: G&O/CNMC-118 dt29.12.2021
Record Dates: First submitted 2022-03-14; First posted 2022-03-31 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Miscarriage
MeSH Terms: conditions — Abortion, Spontaneous | interventions — Mifepristone; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mifepristone (Active Comparator): Participants with 1st trimester miscarriage will receive oral 200mg mifepristone .
  After 48 hours of mifepristone, 800 micro gm misoprostol will be given vaginally for expulsion of product of conception (standard care).
  Interventions: Drug: Mifepristone
- Letrozole (Experimental): Participants with 1st trimester miscarriage will receive 10mg letrozole orally for three consecutive days.
  This is to be followed by tablet misoprostol 800 micro gm vaginally for expulsion of product of conception (standard care).
  Interventions: Drug: Letrozole

INTERVENTIONS:
Drug: Mifepristone — Participants with 1st trimester miscarriage will receive for medical termination
  Other Names: Misoprostol 800 microgram vaginally
  Arms: Mifepristone
Drug: Letrozole — Participants with 1st trimester miscarriage will receive for medical termination
  Other Names: Misoprostol 800 microgram vaginally
  Arms: Letrozole

SUMMARY:
Prospective interventional study where participants with non-viable pregnancy at 1st trimester will be randomized into two arms, one group will receive conventional treatment with oral mifepristone followed by misoprostol vaginally and another group will receive letrozole for three consecutive days followed by misoprostol vaginally in an attempt to terminate the pregnancy medically. Mean duration of induction to expulsion of product of conception and rate of complete abortion will be compared in two groups.

ELIGIBILITY:
INCLUSION CRITERIA :

* Women older than 18years who will give consent regarding medical management of missed abortion
* First trimester pregnancy (gestational age less than equal to 12weeks) with missed abortion confirmed by ultrasonography
* Hemoglobin level more than 12mg/dl

EXCLUSION CRITERIA :

* Hemodynamically unstable patient
* Abnormalities in blood tests including complete blood count (CBC), prothrombin time(PT), internationalised normalized ratio(INR) and fibrinogen
* History or clinical evidence of any thromboembolic impairment or deep venous thrombosis
* Having intra-uterine device
* Present or previous use of corticosteroids
* History of any malignancy
* Existing cardiovascular disease contraindicating misoprostol

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 120 (Estimated)
Dates: Start 2022-05-05 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Expulsion of product of conception | 24 hours since administration of misoprostol
  Mean duration of expulsion since administration of vaginal misoprostol
Requirement of surgical evacuation | beyond 24 hours since misoprostol administration
  Surgical evacuation where complete abortion does not occur

CONTACTS AND LOCATIONS:
Locations (1):
- Calcutta National Medical College and Hospital, Kolkata, West Bengal, India